CLINICAL TRIAL: NCT05869279
Title: Phase I/II Trial to Determine the in Vivo Engraftment, Safety and Clinical Activity of Allogeneic CIK Cells Transduced With a Transposon CD19-chimeric Antigen Receptor (CARCIK-CD19) Gene in Adult and Pediatric Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Allogeneic CARCIK-CD19 in Adults/Pediatric B-cell NHL or Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Matilde Tettamanti Menotti De Marchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT04CARCIK
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-05

CONDITIONS: B-cell NHL; CLL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARCIK-CD19 (Experimental): Gene therapy product composed of T lymphocytes differentiated according CIK-cell protocol (leading to production of CD3+ cells also expressing CD8 and to a lesser extent CD4 or CD56) that have been genetically modified to express CAR with specificity for targeting CD19 molecule expressed on the surface of B cells. The CARCIK-CD19 contains cells that express the anti-CD19 single chain fragment variable (scFV) linked to an intracellular signaling domain comprising the TCR CD3 ζ chain and tandem costimulatory domains as the CD28 and OX40 (CD19-CD28OX40).
  Interventions: Biological: CARCIK-CD19

INTERVENTIONS:
Biological: CARCIK-CD19 — allogeneic cytokine induced killer cells transduced with a transposon CD19-chimeric antigen receptor (CARCIK-CD19) gene

SUMMARY:
This is a single arm, open-label, multi-center, phase I/II study to determine the engraftment, safety and clinical activity of allogeneic CARCIK-CD19 cells in adult and pediatric patients with relapsed/refractory mature B-cell neoplasia expected to express CD19 i.e. B-cell NHL and CLL.

CARCIK-CD19 will be produced from the peripheral blood of an at least haploidentical familial donor.

ELIGIBILITY:
Inclusion Criteria:

criteria apply:

1. Able and willing to provide written informed consent and to comply with the study protocol according to International Conference on Harmonization (ICH) and local regulations.
2. Ineligibility to commercially available CAR-T cells
3. Age limits: children (1-17 years old) and adults (≥18 years old)
4. Availability of an at least haploidentical (i.e. 4/8 HLA matched by allele typing) familial donor willing to and eligible for blood donation
5. Histologically-confirmed mature B-cell neoplasia (NHL), according to according to WHO 2021 classification:

   • Eligible histologies include: indolent [follicular lymphoma (FL) or marginal zone lymphoma (MZL) nodal; extra-nodal; or splenic] or aggressive [diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBL), high-grade B cell lymphoma with MYC and BCL2 rearrangements (double-hit lymphoma), mantle cell lymphoma (MCL), including transformed B-cell NHL], CLL or lymphocytic lymphoma (LL). high-grade B cell lymphoma (HGBCL) NOS. Additional histologies including Burkitt lymphoma and Richter syndrome will be considered upon review with Sponsor.
6. Relapsed after or refractory to at least two prior lines of treatment, and no available treatment options that are expected to prolong survival (e.g. chemotherapy or high-dose chemotherapy/stem cell transplantation, commercially available CART cell therapy or other standard treatment) or patients refusing such treatments
7. At least one measurable target lesion, measurable as defined by Lugano 2014 classification (nodal: > 1.5 cm longest transverse diameter; extra-nodal: > 1 cm longest transverse diameter) by computerized tomography (CT) scan or presence of assessable disease (i.e. bone marrow or spleen)
8. Eastern Cooperative Oncology Group (ECOG) performance status equal to 2 or less for subject ≥ 16 years of age, or Lansky >50 for subjects < 16 years of age
9. Adequate cardiac and pulmonary function: ejection fraction (EF) by echo or MUGA >40% and radial artery (RA) oxygen saturation >92%.
10. Life expectancy (in the opinion of the Investigator) of > 12 weeks
11. Adequate liver function:

    * Total bilirubin ≤ 2.0x ULN (≤ 3x ULN in patients with Gilbert's syndrome or documented liver involvement)
    * AST (aspartate aminotransferase) /ALT (alanine aminotransferase) 3x ULN or 5x for patients with evidence of liver involvement with lymphoma
12. Adequate bone marrow function to receive lymphodepleting chemotherapy at investigator judgment.
13. Adequate renal function: creatinine ≤1.5x ULN or creatinine clearance (CrCl) calculated by Cockcroft-Gault formula of ≥50 mL/min for adult patients in whom, in the Investigator's judgment, serum creatinine levels do not adequately reflect renal function. For children, CrCl will be calculated by local institutional standard.
14. Females of childbearing potential (FCBP) subjects must:

    * Have a negative pregnancy test as verified by the local investigator
    * Either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption from screening until at least 12 months following CARCIK-CD19 infusion and until CAR positive viable T cells are no longer present by quantitative polymerase chain reaction (qPCR) on two consecutive tests.
    * Contraception methods must include one highly effective method including: surgical female sterilization, use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%)
    * Agree to abstain from breastfeeding during study participation and for at least 12 months following CARCIK-CD19 infusion and until CAR positive viable T cells are no longer present by quantitative polymerase chain reaction (qPCR) on two consecutive tests.
15. Male subjects must:

    * Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential for 12 months after following CARCIK-CD19 infusion and until CAR positive viable T cells are no longer present by quantitative polymerase chain reaction (qPCR) on two consecutive tests.

Exclusion Criteria:

1. Patients with clinically significant active viral, bacterial or fungal infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 2 weeks prior to CARCIK-CD19 infusion.
2. Patients with an active infection with Hepatitis B. However, patients with a controlled (treated) hepatitis will be allowed if the all the following criteria are met:

   * Anti-viral therapy for hepatitis B virus (HBV) must be given for at least 1 month prior to time of informed consent;
   * HBV viral load must be <2000 IU/mL (104 copies/mL) prior to time of informed consent; and
   * those on active HBV therapy with viral load <2000 IU/mL (104 copies/mL) should stay on the same anti-viral therapy throughout study treatment
3. Patients with an active hepatitis C virus (HCV) infection. However, patients with successfully treated chronic HCV infection will be allowed if they show a sustained virologic response at 12 weeks (SVR12) or 24 weeks (SVR24), and if there is a 4-week period between achieving sustained viral response (SVR12 or SVR24) and time of informed consent.
4. Patients with a positive serologic test or a positive molecular PCR test for human immunodeficiency virus (HIV) are eligible if asymptomatic, well controlled by the HAART therapy and no medically significant active infection is present
5. Rapidly progressive disease that in the estimation of the investigator and sponsor could affect compliance with the protocol or interpretation of results
6. Active CNS lymphoma
7. Major surgery or significant traumatic injury 28 days prior to CARCIK-CD19 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
8. Patients with another active invasive malignancy with a life expectancy of less than 3 years
9. Significant cardiovascular disease (such as New York Heart Association (NYHA) Class II cardiac disease, congestive heart failure, myocardial infarction or cerebrovascular accident within 30 days prior to CARCIK-CD19 infusion, unstable arrhythmias, or unstable angina)
10. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders (bronchospasm, obstructive pulmonary disease) and known autoimmune diseases
11. Treatment with any other standard anti-cancer radiotherapy / chemotherapy including investigational therapy (defined as treatment for which there is currently no regulatory authority approved indication) within 2 weeks prior to CARCIK-CD19 infusion
12. Allogeneic or autologous Stem Cell Transplantation within 3 months prior to CARCIK-CD19 infusion, or Donor Lymphocytes (DLI)
13. Active GvHD Grades II-IV or extensive chronic Graft-versus-Host Disease (for patients who had previously been allotransplanted)
14. Prior treatment with CART cell therapy within 30 days before first study treatment administration (lymphodepletion)
15. Toxicities from prior anti-cancer therapy including immunotherapy that did not resolve to ≤ Grade 1 with the exception of alopecia, endocrinopathy managed with replacement therapy and stable vitiligo.
16. Ongoing corticosteroid use 25 mg/day (> or 0.3 mg/kg for children) of prednisone or equivalent within 1 weeks prior to CARCIK-CD19 infusion
17. Administration of a live, attenuated vaccine within 4 weeks prior to CARCIK-CD19 infusion

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 day after CARCIK infusion
  Dose Limiting Toxicity
overall response rate | month 3 after CARCIK-CD19 infusion
  overall response rate (complete + partial remission)

SECONDARY OUTCOMES:
Adverse event (AE) | up to 12 months
  Incidence of Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Biondi, MD, Principal Investigator — IRCCS San Gerardo dei Tintori
Locations (1):
- Ospedale Papa Giovanni XXIII, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No